CLINICAL TRIAL: NCT03284047
Title: Evaluation of Different Doses of Botulinum Toxin Type A for the Treatment of Gummy Smile
Brief Title: Botox for Gummy Smile
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00205065
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Gingival Exposure
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2.5 U dose (Experimental): Participants with more than 4 mm of upper anterior gingival exposure measured from the central incisor tooth will be randomly assigned (1:1:1) to receive different doses of botulinum toxin type A (abobotulinumtoxin A) on the levator labii superioris alaeque nasi as follows:
  1. 2.5 U
  2. 5 U
  3. 7.5 U
  Interventions: Drug: Botulinum toxin type A
- 5 U dose (Experimental): Participants with more than 4 mm of upper anterior gingival exposure measured from the central incisor tooth will be randomly assigned (1:1:1) to receive different doses of botulinum toxin type A (abobotulinumtoxin A) on the levator labii superioris alaeque nasi as follows:
  1. 2.5 U
  2. 5 U
  3. 7.5 U
  Interventions: Drug: Botulinum toxin type A
- 7.5 U dose (Experimental): Participants with more than 4 mm of upper anterior gingival exposure measured from the central incisor tooth will be randomly assigned (1:1:1) to receive different doses of botulinum toxin type A (abobotulinumtoxin A) on the levator labii superioris alaeque nasi as follows:
  1. 2.5 U
  2. 5 U
  3. 7.5 U
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Participants will be randomized to one of three botulinum toxin type A doses.

SUMMARY:
This is a two part study to measure and observe the efficacy of botulinum toxin A for the treatment of gummy smiles.

Part A will randomly compare three different doses of botulinum toxin type A (abobotulinumtoxin A) for the treatment of upper anterior gummy smile with larger gingival exposure (> 4 mm).

Part B will assign one of two doses of botulinum toxin type A for participants with smaller gingival exposure (< 4 mm).

Follow-up visits with photography will occur 4 and 12 weeks after their treatment. Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

This study is a pilot study designed to determine feasibility of this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Males or females ≥ 18 years old
3. Anterior gingival exposure during smiling larger than 4 mm measured from the central incisor tooth (part A), or 2-4 mm (part B).
4. Subjects of childbearing potential who present a negative urine pregnancy test at baseline and use an effective contraceptive method.
5. Subjects are in good health as judged by the investigator.
6. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

1. Pregnant women or women intending to become pregnant in the next 8 months after the screening for eligibility
2. Subjects participating in other clinical trials
3. Any prior surgery affecting the area of study
4. Subjects with neoplastic, muscular or neurological disease
5. Subjects who have received botulinum toxin treatment for gummy smile in the previous 12 months before the inclusion date
6. Subjects who have received Botulinum toxin treatment for any other cosmetic indication in the previous 6 months before the inclusion date
7. Subjects using aminoglycosides and penicillamine antibiotics, quinine or calcium channel blockers
8. Subjects with inflammation or active infection in the area to be injected
9. Subjects with history of sensitivity to the components of the formulation.
10. Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
11. Subjects who are unable to understand the protocol or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-24 (Estimated); Primary Completion 2019-04-24 (Estimated); Study Completion 2019-04-24 (Estimated)

PRIMARY OUTCOMES:
Reduction of the upper gum exposure at 4 weeks and 12 weeks. | [Baseline, 4 weeks,12 weeks]
  Reduction in millimeters in the upper gum exposure of subjects after botulinum toxin type A (abobotulinumtoxin A) treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No